CLINICAL TRIAL: NCT02974244
Title: A Cohort Study of the Benefits of Bydureon in Customary Clinical Care in the United States
Brief Title: Comparison of the Effectiveness and Tolerability of Exenatide Once-weekly Compared to Basal Insulins
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5551R00008
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- exenatide once weekly: type 2 diabetes who initiated exenatide once weekly treatment in the index period
  Interventions: Drug: exenatide once weekly
- basal insulin: type 2 diabetes patients who initiated basal insulin treatment in the index period
  Interventions: Drug: basal insulin

INTERVENTIONS:
Drug: exenatide once weekly — exenatide treatment in the customary clinical care in the USA
  Groups: exenatide once weekly
Drug: basal insulin — basal insulin treatment in the customary clinical care in USA
  Groups: basal insulin

SUMMARY:
Exenatide once weekly (Bydureon) was approved in January 2012 by FDA in USA for the treatment of type 2 diabetes mellitus. Evidence from clinical trials suggested that Bydureon improves glucose control with low risk of hypoglycemia. Bydureon does not require a dose titration as necessary for other glucagon-like peptide-1 agonists, and appears to have other advantages, such as reducing insulin resistance, reducing weight, and improving blood pressure and lipid profiles. However, the degree to which these advantages of Bydureon lead to improve outcomes in customary clinical care is unknown.

The aim of this study is to evaluate the effectiveness and tolerability of Bydureon relative to basal insulin initiated as first-ever injectable therapeutic regimens used in customary clinical care. Patients who initiated treatment with Bydureon or basal insulin between July 2011 and March 2015 will be recruited into the study cohorts from Optum's database of electronic health records. The two treatment cohorts will be matched by propensity score method.Clinical outcomes of HbA1c, weight, and gastrointestinal symptoms and hypoglycemia are investigated.

DETAILED DESCRIPTION:
Background: In January 2012, the US Food and Drug Administration approved a once-weekly form of exenatide, Bydureon, for the treatment of type 2 diabetes mellitus. Evidence from clinical trials suggested that Bydureon improves glucose control with low risk of hypoglycemia. Bydureon does not require a dose titration as necessary for other glucagon-like peptide-1 receptor agonists (GLP-1RAs), and appears to have other advantages, such as reducing insulin resistance, preventing weight gain, and improving blood pressure and lipid profiles. However, the degree to which these advantages of Bydureon lead to improve outcomes in customary clinical care is unknown.

Aims: The aim of this study is to evaluate the effectiveness and tolerability of Bydureon relative to basal insulin initiated as first-ever injectable therapeutic regimens used in customary clinical care.

The specific study objectives are as follows:

* To quantify the effectiveness of Bydureon initiation relative to initiation of basal insulin, on improving:
* Glycated hemoglobin (HbA1c)
* Weight (body mass index (BMI))
* HbA1c simultaneous to reduction in weight
* Blood pressure and lipid profiles
* To monitor the tolerability of Bydureon initiation relative to initiation basal insulin, on the occurrence of :
* Hypoglycemia
* Gastrointestinal symptoms (nausea, vomiting, diarrhea, and constipation)
* Change in the markers for renal disease (estimated glomerular filtration rate (eGFR), serum creatinine, and albumin/creatinine ratio (ACR), and the stability of liver function test (AST, ALT) and standard blood counts (white blood cell, red blood cell, Hematocrit, Hemoglobin, Platelet)
* To examine these measures of effectiveness and tolerability within potentially vulnerable subgroups of Bydureon and basal insulin initiators:
* Type 2 diabetes patients with renal impairment
* Elderly Type 2 diabetes patients
* Type 2 diabetes patients who are a minority race
* Type 2 diabetes patients within strata of HBA1c Design: This retrospective cohort study will be conducted using Optum's electronic health record data from July 2011 through March 2015 and identified injectable-naive Type 2 diabetes patients who initiated either Bydureon or basal insulin during the accrual period, January 2012 and January 2015. Injectable-naive Type 2 diabetes patients will be identified. Propensity score methods will be used to match initiators of Bydureon to basal insulin initiators.

Study Population:

The study population will be selected from the electronic health recrod data included patients with Type 2 diabetes who initiated Bydureon or basal insulin. Eligible patients had:

* Received care for at least 6 months prior to the date of study drug initiation (cohort entry) with at least one outpatient clinic visit in the 6 months prior to cohort entry (baseline period);
* At least one diagnosis of type 2 diabetes (ICD-9 250.X0 or 250.X2) prior to and including the date of the qualifying drug initiation, no prior diagnosis (inclusive of the index date) of type 1 diabetes mellitus (250.X1 or 250.X3), and no diagnosis of gestational diabetes within the previous 6 months (inclusive of the index date); and
* No evidence of prior injectable antidiabetic treatment, specifically no dispensing of GLP-1RA or any insulin drug during the 6-month baseline period. Outcomes and Analysis: To measure the effectiveness of Bydureon relative to basal insulin are changes in HbA1c and body weight, as well as changes in HbA1c and simultaneous reduction in weight. Changes in BMI, lipid profiles, and blood pressure will be examined. These variables are part of the clinical and laboratory data in the electronic health records. Each outcome will be evaluated for completeness, multiply imputed, and reported across standardized time intervals. HbA1c, weight and BMI are summarized in baseline and quarterly (3-month intervals) in the first year following drug initiation. Lipid measurements and blood pressure are summarized in baseline and bi-annually (6-month intervals) in the first year following drug initiation.

To assess drug tolerability, the incidence of hypoglycemia, and gastrointestinal symptoms (nausea, vomiting, diarrhea, and constipation) will be assessed. These outcomes are ascertained using an ICD-9 algorithm applied to the structured fields and by extracting mentions of hypoglycemia using a natural language processing (NLP) algorithm developed by Optum and applied to the free text clinical notes available in the data. In addition the stability of renal function evaluated by change in eGFR, or albumin/creatinine ratio (ACR); the change in serum hepatic enzymes [aspartate aminotransferase (AST), alanine aminotransferase (ALT)], and hematologic measures [red blood cells counts (RBC), white blood cell counts (WBC), platelets (PLT), hemoglobin (Hgb) and hematocrit (Hct) will be evaluated. Each of these laboratory values will be evaluated for completeness, multiply imputed, and reported across standardized time intervals. eGFR and ACR will be summarized in baseline and quarterly (3-month intervals) in the first year following drug initiation. Hepatic enzymes and hematologic measures are summarized in baseline and semi-annually (6-month intervals) in the first year following drug initiation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* had received care documented in Electronic Health Records (including at least one out-patient provider visit) for a minimum of 6-months prior index date;
* had at least one diagnosis of type 2 diabetes by The International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM: 250.X0 or 250.X2) prior to and including the date of the study drug initiation, with no prior diagnosis of type1 diabetes (ICD-9-CM: 250.X1 or 250.X3), or gestational diabetes within the 6-months prior to index date;
* No evidence of prior injectable antidiabetic treatment, specifically no dispensing of a GLP-1RA or any insulin during the 6-months baseline period prior to study drug initiation

Exclusion Criteria:

* Prior diagnosis of type1 diabetes (ICD-9-CM: 250.X1 or 250.X3), or gestational diabetes within the 6-months prior to index date;
* Prior dispensing of a GLP-1RA or any insulin

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study compares injectable-naive exenatide once-weekly and basal insulin initiators. The study cohorts were drawn from an Optum's Electronic Health Records database that integrates records from many medical groups and hospitals in the United States representing over 25,000 physicians and over 25 million patients in ordinary clinical practice. The Electronic Health Records captures clinical, operational, and financial information that physicians record at the time of care. This information includes diagnoses, procedures, medications (prescribed and administered), clinical measures (biometric and laboratory values), and clinical notes (e.g., physician, pathology, and radiology notes).
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2014-10-28 (Actual); Study Completion 2014-10-28 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in HbA1c (%) | one year post-index
  To evaluate changes in HbA1c from baseline one year after starting treatment with exenatide once weekly and basal insulin
Changes from baseline in weight (kg) | one year post-index
  To evaluate changes in weight (kg) from baseline one year after starting treatment with exenatide once weekly and basal insulin

SECONDARY OUTCOMES:
Frequency of hypoglycemia | one year post-index
  to evaluate frequency of hypoglycemia in association with initiation of therapy with exenatide once weekly and basal insulin
Frequency of nausea | One year post-index
  to evaluate frequency of nausea in association with initiation of therapy with exenatide once weekly and basal insulin
Frequency of vomiting | one year post-index
  to evaluate frequency of vomiting in association with initiation of therapy with exenatide once weekly and basal insulin
Frequency of diarrhea and constipation | One year post-index
  to evaluate frequency of diarrhea and constipation in association with initiation of therapy with exenatide once weekly and basal insulin

CONTACTS AND LOCATIONS:
Overall Officials: Anita M Loughlin, Ph.D, Principal Investigator — Optum, Inc.
Locations (1):
- Optum Epidemiology, Boston, Massachusetts, United States

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4433&filename=D5551R00008_Poster_ADA2016.pdf